CLINICAL TRIAL: NCT03877770
Title: Is Deep Vein Thrombosis an Under-recognised Complication of Electrophysiology Procedures? A Mechanistic Observational Study Investigating Markers and Incidence of Thromboembolism
Brief Title: DVT After Cardiac Procedure
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 219270
Record Dates: First submitted 2019-02-15; First posted 2019-03-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Thromboembolism; Deep Vein Thrombosis
MeSH Terms: conditions — Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients undergoing electrophysiology studies (EPS) and cardiac ablation procedure for the treatment of cardiac arrhythmias may be at increased risk of deep vein thrombosis (DVT) during or after the procedure, which may lead to pulmonary embolus which can be life threatening. The study will use Doppler ultrasound scanning at 24h and between 10-14 days post EPS and cardiac ablation to assess the incidence of undiagnosed DVT. A positive finding may provide support for a larger clinical trial to assess the benefit of prophylactic anticoagulation post EPS procedure.

DETAILED DESCRIPTION:
Electrophysiological study (EPS) and catheter ablation is an established method for the assessment and treatment of many patients with cardiac arrhythmias (altered heart rhythm). It is generally carried out in patients who are usually otherwise fairly fit and healthy. In the UK many patients undergo this procedure and the numbers are increasing. The procedure involves a number of catheters (tubes) being inserted into the femoral vein over a period of up to 2 ½ hours. Presence of the catheter in the vein increases the risk of blood clot formation, if a clot blocks a deep vein in the leg (deep vein thrombosis), it can lead to pain and chronic leg swelling as well as the need for blood thinning (anticoagulant) medications. In some patients, fragments of the blood clot can break off and travel to the lungs which can be life-threatening. It is important to detect the presence of a clot as soon as possible, so that treatment may be given. The investigators hope to establish if the condition is more common than originally thought.

The investigators plan to recruit 100 patients who are due to undergo EPS or catheter ablation. Prior to the participant's clinical procedure, the investigators will perform an additional blood test to check blood clotting function. After the cardiac procedure, the participants will then undergo Doppler ultrasound scans at 24 hours and a second scan between 10-14 days to check for the presence of blood clots.

The aim of the study is to increase understanding of how often these blood clots occur and confirm if blood tests or current gold-standard imaging is best at showing the early stages of blood clot formation. The results of the study will help decide if a clinical trial is needed to test whether giving preventative blood thinning treatment after cardiac procedures would be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 80 undergoing elective EP study and catheter ablation
* Procedure duration between 30 minutes - 4 hours from the time of venous puncture to sheath removal
* 3-5 sheaths in a femoral vein

Exclusion Criteria (pre-procedure):

* Under 18
* Electrophysiology study only (no ablation performed)
* Inadequate understanding of spoken English
* Intubated/ventilated patients
* Unwilling to give consent to participation OR advised by consultee that this would be against the patient's wishes.
* Recently treated infection
* Intravascular implanted cardiac device
* Prior pacemaker extraction
* Prior cardiac surgery
* Previous cardiac ablation within 6 months
* Documented atrial flutter or atrial fibrillation within 1 year prior to ablation procedure.
* Participation in a clinical trial of an investigational medicinal product (CTIMP)
* Documented previous venous thrombosis or pulmonary embolism
* Known coagulopathy or anticoagulant use
* Known use of anti-platelet agent
* Known concurrent clinical problem likely to interfere with participation or completion of the study

Exclusion criteria (post-procedure):

* EPS carried out without ablation
* Left sided ablation or other clinical mandate for perioperative anticoagulation
* Complications during procedure (including arterial puncture or failure to advance venous wires)
* Peri-procedural complications that would, in the opinion of the PI/designee preclude further participation in the study
* Post-procedure bleeding or haematoma formation requiring prolonged (>30 minutes) pressure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for elective EP study and catheter ablation.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Presence of DVT as evidenced by Doppler Ultrasound | Up to 14 days post procedure.
  The incidence of DVT in the treated leg will be reported. The study will use Doppler ultrasound scanning post EPS and cardiac ablation to assess the incidence of undiagnosed DVT at up to 14 days post procedure.

SECONDARY OUTCOMES:
Elevation of blood markers of DVT in the absence of clinically detectable DVT. | Blood sampling takes place pre-ablation and 24 hours post procedure.
  The d-dimer blood sample is taken as part of the research assessment to determine its use as a marker of thrombus formation following invasive procedure.The outcome would be to see if more significant elevation is seen in patients with thrombus and whether a baseline elevated level would put you at higher risk of thrombus.
Ultrasound characteristics of the DVT, and change between scans. | Up to 14 days post procedure.
  The study will use Doppler ultrasound scanning post EPS and cardiac ablation to assess the incidence of undiagnosed DVT at up to 14 days post procedure.
The occurrence of DVT in the untreated leg. | Up to 14 days post procedure.
  The DVT incidence in the treated leg will be compared to both that in the control leg and known background incidence from the literature.The study will use Doppler ultrasound scanning post EPS and cardiac ablation to assess the incidence of undiagnosed DVT at up to 14 days post procedure.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, Lancashire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, Yorkshire
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruce C, Saraf K, Rogers S, El-Omar M, Kirkwood G, Kelland NF, Shah D, Chalil S, Fullwood C, Wright M, Jamil-Copley S, Fox D, Abozguia K, Thachil J, McCollum C, Morris GM. Deep Vein Thrombosis is Common After Cardiac Ablation and Pre-Procedural D-Dimer Could Predict Risk. Heart Lung Circ. 2022 Jul;31(7):1015-1022. doi: 10.1016/j.hlc.2022.01.014. Epub 2022 Mar 14. PMID 35301985